CLINICAL TRIAL: NCT03603756
Title: SHR-1210, a Novel Anti-PD-1 Antibody, in Combination With Apatinib and Irinotecan/Paclitaxel Liposome Plus Nedaplatin in Patients With Previously Untreated Advanced or Metastatic Esophageal Squamous Cell Cancer: a Phase II Study
Brief Title: SHR-1210 in Combination With Apatinib and Chemotherapy in Patients With Advanced Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC201807010
Record Dates: First submitted 2018-07-20; First posted 2018-07-27 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; apatinib; Irinotecan; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients with advanced or metastatic esophageal squamous cell carcinoma are to receive SHR-1210 with apatinib and irinotecan injection in cohort 1.
  Interventions: Drug: SHR-1210; Drug: Apatinib; Drug: Irinotecan Injection
- Cohort 2 (Experimental): Patients with advanced or metastatic esophageal squamous cell carcinoma are to receive SHR-1210 with apatinib and paclitaxel liposome plus nedaplatin in cohort 2.
  Interventions: Drug: SHR-1210; Drug: Apatinib; Drug: Paclitaxel liposome; Drug: Nedaplatin

INTERVENTIONS:
Drug: SHR-1210 — a novel anti-PD-1 antibody
Drug: Apatinib — a VEGFR-2 tyrosine kinase inhibitor
Drug: Irinotecan Injection — cytotoxic agent that binds to topoisomerase I
  Arms: Cohort 1
Drug: Paclitaxel liposome — cytotoxic agent that prevent depolymerization of cellular microtubules
  Arms: Cohort 2
Drug: Nedaplatin — cytotoxic agent that cross-links and denatures strands of DNA
  Arms: Cohort 2

SUMMARY:
Patients with previously untreated advanced or metastatic esophageal squamous cell carcinoma are recruited to this prospective non-randomized study comprising two separate cohorts. Patients will receive SHR-1210, a novel anti-PD-1 antibody, with apatinib and either irinotecan or paclitaxel liposome plus nedaplatin. The primary endpoint is to determine the objective response rate (ORR) of patients in both cohorts. The regimen(s) of promising efficacy will be further verified in subsequent randomized studies to define the optimal combination of immunotherapy, anti-angiogenesis and chemotherapy in advanced esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell carcinoma of the esophagus, locally advanced, unresectable, recurrent or metastatic disease.
2. Have not received prior systemic therapy.
3. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
4. Eastern Collaborative Oncology Group (ECOG) Performance Status ≤ 1.
5. Life expectancy >12 weeks.
6. Adequate organ function.
7. For females of child bearing potential, a negative urine or serum pregnancy test result within 72h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study until 2 months after the last dose of any of the drugs in the study.
8. Willing and able to provide written informed consent and comply with the requirements of the study.

Exclusion Criteria:

1. Any previous malignancy, except for non squamous-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix within 5 years prior to study entry.
2. Known central nervous system (CNS) metastases.
3. Prior therapy with any of the immune check-point inhibitors.
4. Known immediate or delayed hypersensitivity reaction to SHR-1210, apatinib, irinotecan, paclitaxel liposome, nedaplatin or their excipients.
5. Subjects with any active autoimmune disease or history of autoimmune disease.
6. Known Human Immunodeficiency Virus (HIV) infection, active Hepatitis B or Hepatitis C infection.
7. Concurrent medical condition requiring the use of cortisol (>10mg/day prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids no more than 10 mg/day prednisone or equivalent.
8. Received a live vaccine within 4 weeks of the first dose of study medication.
9. Hypertension with a blood pressure of systolic> 140 millimeter of mercury (mm Hg) and/or diastolic > 90 mm Hg that is not effectively controlled by anti-hypertensive therapy.
10. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention.
11. Unable to swallow oral medications or with gastrointestinal disorders that might interfere with proper absorption of oral drugs.
12. Active digestive ulcer disease, inflammatory bowel disease, intestinal obstruction or any other condition that, in the clinical judgment of the Principal Investigator, may cause severe gastrointestinal bleeding or perforation.
13. Active infection or an unexplained fever > 38.5°C before 4 weeks of enrollment.
14. Unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolic conditions.
15. Pregnant or lactating female.
16. Familial, sociological or geographical conditions that, in the clinical judgment of the Principal Investigator, do not permit compliance with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-03-28 (Estimated); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 24 months
  objective response rate of the patients in cohort 1 and cohort 2

SECONDARY OUTCOMES:
progression-free survival (PFS) | 24 months
  progression-free survival (PFS) of the patients in cohort 1 and cohort 2
overall survival | 24 months
  overall survival of the patients in cohort 1 and cohort 2
treatment-related adverse events | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Principal Investigator — Cancer Hospital,CAMS
Locations (1):
- Jing Huang, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang B, Qi L, Wang X, Xu J, Liu Y, Mu L, Wang X, Bai L, Huang J. Phase II clinical trial using camrelizumab combined with apatinib and chemotherapy as the first-line treatment of advanced esophageal squamous cell carcinoma. Cancer Commun (Lond). 2020 Dec;40(12):711-720. doi: 10.1002/cac2.12119. Epub 2020 Dec 12. PMID 33314747